CLINICAL TRIAL: NCT07231718
Title: The Effectiveness of an AI-Supported Cyberbullying Awareness Program on Adolescents' Cyberbullying: A Randomized Controlled Trial
Brief Title: The Effectiveness of an AI-Supported Cyberbullying Awareness Program on Adolescents' Cyberbullying
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: M. Furkan Kurnaz (Other)
Responsible Party: Sponsor-Investigator, M. Furkan Kurnaz, Assistant Professor, Necmettin Erbakan University
Organization: Necmettin Erbakan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEU27674
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: AI-supported Cyberbullying Awareness Program

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist (No Intervention): Adolescents in waitlist group will not receive AI-supported cyberbullying awareness program.
- Experimental Group (Experimental): The cyberbullying awareness program with AI-supported videos
  Interventions: Other: AI-supported cyberbullying awareness program.

INTERVENTIONS:
Other: AI-supported cyberbullying awareness program. — Participants in this arm will receive the Ministry of National Education's (MEB) cyberbullying awareness program, supplemented with AI-supported instructional videos. The intervention includes standard psychoeducational materials developed by MEB and UNICEF, along with digital videos that use AI to personalize feedback, provide scenario-based learning, and guide students through interactive exercises related to recognizing, preventing, and responding to cyberbullying. Delivery occurs through sessions in which participants watch AI-supported instructional videos integrated into the standard MEB cyberbullying awareness program.
  Arms: Experimental Group

SUMMARY:
With the increasing prevalence of cyberbullying among adolescents today, there is a greater focus on interventions targeting cyberbullying. In Turkey, cyberbullying awareness programs developed in collaboration between the Ministry of National Education (MEB) Directorate General of Special Education and Guidance Services and the United Nations Children's Fund (UNICEF) are being used. This study aims to examine the effectiveness of the cyberbullying awareness program developed by the MEB by enriching it with AI-supported content.

DETAILED DESCRIPTION:
With the advancement of technology, most adolescents can easily access online environments for various purposes such as communicating with others, playing games, searching for information, and socializing. Although this development offers adolescents many opportunities, it can also cause them to encounter some difficult situations. One of these difficulties is cyberbullying, which adolescents encounter in online environments. This research is important because it aims to increase adolescents' awareness of cyberbullying and examine the reduction of cyberbullying behaviors among adolescents using an awareness program enriched with AI-supported content.

ELIGIBILITY:
Inclusion Criteria:

* the study include being an adolescent.

Exclusion Criteria:

* Not having any specific mental health disorder.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Revised Cyber Bullying Inventory-II (RCBI-II) | baseline, within 1 minute after the fourth session, within 1 minute post-test, and 3 months follow-up
  The Revised Cyberbullying Inventory-II (RCBI-II), revised by Topçu and Erdur-Baker (2017), assesses the levels of cyberbullying behaviors among adolescents. The RCBI-II consists of two forms: cyberbullying perpetration and cyberbullying victimization, with each form comprising 10 items. Items are rated on a four-point scale ranging from 1 (It has never happened to me) to 4 (It happened more than five times). High scores on the forms indicate high levels of cyberbullying victimization and perpetration.

CONTACTS AND LOCATIONS:
Overall Officials: M. Furkan Kurnaz, PhD, Study Chair — Necmettin Erbakan University
Locations (1):
- Eregli High School Education, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No